CLINICAL TRIAL: NCT03732781
Title: A Phase 1/2a Study to Evaluate the Dose, Safety and Tolerability and Efficacy of an Intraperitoneal α-emitting Radionuclide Therapy (Radspherin®) in Subjects With Peritoneal Carcinomatosis From Colorectal Carcinoma Following Hyperthermic Intraperitoneal Chemotherapy
Brief Title: Study of Radspherin® in Colorectal Carcinoma Subjects With Peritoneal Carcinomatosis Treated With HIPEC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oncoinvent AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RAD-18-002; 2018-002803-33 (EudraCT Number)
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Peritoneal Carcinoma; Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: 3+3 Dose escalation with expansion cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radspherin (Experimental)
  Interventions: Drug: Radspherin

INTERVENTIONS:
Drug: Radspherin — Radspherin® suspension consists of degradable calcium carbonate microparticles with the α-emitting radionuclide 224Ra in suspension.
  Radspherin® will be provided in a R10 vial filled with 10 mL suspension of 224Ra adsorbed on 1 g calcium carbonate microparticles. The volume to be administered will contain 0.7-1 g calcium carbonate microparticles with 1-7 MBq 224Ra. 224Ra has a half-life of 3.6 days.

SUMMARY:
This is a phase 1/2a open label study to evaluate the dose, safety, tolerability and efficacy of an IP α-emitting radionuclide therapy (Radspherin®) in subjects with peritoneal carcinomatosis (PC) from colorectal carcinoma following complete CRS (cytoreduction score CC-0) and HIPEC.

The study consists of three different cohorts:

* Dose escalation cohorts
* Repeated injection cohorts
* Expansion cohort

DETAILED DESCRIPTION:
Primary objectives:

* To investigate safety and toxicity of Radspherin®
* To determine the maximum-tolerated dose (MTD) of Radspherin®, among the four suggested doses 1, 2, 4 and 7 MBq, as a single intraperitoneal (IP) injection and two repeated IP injections following cytoreductive surgery (CRS) and hyperthermic IP chemotherapy (HIPEC)

Secondary objectives:

* To establish a recommended dose of Radspherin® as a single IP injection and two repeated IP injections following CRS and HIPEC
* To describe the biodistribution of Radspherin®
* To examine the efficacy and clinical benefit of Radspherin® following CRS and HIPEC

Exploratory objectives:

* To explore the association of biomarkers with activity/clinical benefits, adverse events (AEs), or other effects associated with Radspherin®
* To explore effects of catheter placement, Radspherin® administration technique, and infusion volume on the distribution of 224Ra labelled micro particles in the peritoneal cavity

The maximum number of subjects receiving Radspherin® in this study is 67. Subjects who discontinue prior to Radspherin® administration will be replaced.

Dose escalation cohorts: 3 - 24 subjects Repeated injection cohorts: 3 subjects Expansion cohort: up to 40 subjects

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent and to comply with the clinical study protocol
2. Age ≥ 18 years
3. Histologically confirmed colorectal carcinoma
4. Peritoneal metastases (PCI≤20 assessed during surgery), and histologically confirmed as peritoneal carcinomatosis) eligible for cytoreductive surgery and HIPEC treatment that reaches CC-0 at the end of the surgical procedure
5. AEs recovered to at least grade 1 from the effects (excluding alopecia) of any prior medical therapy for malignancy at time of first administration of Radspherin®
6. ECOG Performance Status Score of 0 - 1
7. Adequate renal function

   * Creatinine ≤ 1.8 mg/dl (159 μmol/l) and
   * Calculated creatinine clearance using the Cockcroft-Gault formula ≥ 45 ml/min, or
   * Measured creatinine clearance ≥ 45 ml/min
8. Adequate hepatic function

   * Serum bilirubin <1.5 x upper limit of normal (ULN)
   * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 x ULN
9. Adequate bone marrow function:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/l
   * Platelets ≥ 100 x 109/l
   * Haemoglobin ≥ 9 g/dL
10. Adequate coagulation tests: INR ≤ 1.5 x ULN
11. For females of childbearing potential, a negative pregnancy test must be documented prior to enrolment
12. For females of childbearing potential; agreement to use at least one of the following highly effective (failure rate<1%) methods of contraception during the treatment period and for at least 12 months after the last dose of IMP:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject), periodic abstinence (e.g.: calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before enrolment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment
    * Male sterilization (at least 6 months prior to enrolment). The vasectomized male partner should be the sole partner of the subject
    * Use of oral, (estrogen and progesterone), injected or implanted hormonal methods of contraception or placement of an IUD or IUS, or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception. In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
13. For non-sterile males who's female partner is of childbearing potential: agreement to use condom during the treatment period and for at least 12 months after the last dose of investigational medicinal product. The female partner should use at least one of the following highly effective (failure rate<1%) methods of contraception during the treatment period and for at least 12 months after the last dose of the investigational medicinal product (IMP):

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject), periodic abstinence (e.g.: calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before enrolment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment
    * Use of oral, (estrogen and progesterone), injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception. In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

Note: Male sterilization must have been performed at least 6 months prior to enrolment. A condom is required for all sexually active male subjects during the treatment period and for at least 12 months after the last dose.

• Agree to refrain from donating sperm for the entire treatment period and for up to 12 months after the last dose.

Exclusion Criteria:

1. Peritoneal metastasis originating from appendix vermiformis. Other synchronous visceral metastatic lesions in liver or lungs, symptomatic central nervous system (CNS) metastases. Metastatic lymph nodes or thoracic lymph nodes
2. Resection or suture of the diaphragm (assessed during surgery)
3. Pregnant or lactating (nursing) women
4. Active infections requiring antibiotics and/or physician monitoring, or recurrent fever >38.0⁰C associated with a clinical diagnosis of active infection
5. Active liver disease with positive serology for active hepatitis B, hepatitis C or known HIV
6. Administration of an investigational medicinal product within 28 days or at least 5 times the half-life
7. Concurrent administration of any other cancer therapy other within 4 weeks prior to, and up to 4 weeks after the last study treatment
8. Another primary malignancy within the past 3 years (except for non-melanoma skin cancer, cervical cancer in situ or in situ stage 1 synchronous endometrial cancer)
9. Concurrent congestive heart failure or prior history of New York Heart Association (NYHA) class III/IV cardiac disease
10. Any condition or illness that, in the opinion of the Investigator or the medical monitor, would compromise the safety of the subjects or interfere with the evaluation of the safety of the IMP
11. In the Investigator's opinion not able to comply with study procedures. Any medical or psychological condition that would preclude participation in the study or compromise the ability to give informed consent
12. Known hypersensitivity to any of the excipients in the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicities as assessed by CTCAE v5.0. | 18 months
  To investigate safety and toxicity of Radspherin®
Maximum Tolerated Dose | 21 Days
  To determine the maximum-tolerated dose (MTD) of Radspherin®, among the four suggested doses 1, 2, 4 and 7 MBq, as a single intraperitoneal (IP) injection and two repeated IP injections following cytoreductive surgery (CRS) and hyperthermic IP chemotherapy (HIPEC)
Explore efficacy (expansion cohort) | 18 months
  Peritoneal recurrence free survival

CONTACTS AND LOCATIONS:
Locations (2):
- Oslo University Hospital, Oslo, Norway
- Akademiska, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Larsen SG, Graf W, Mariathasan AB, Sorensen O, Spasojevic M, Goscinski MA, Selboe S, Lundstrom N, Holtermann A, Revheim ME, Bruland OS. First experience with 224Radium-labeled microparticles (Radspherin(R)) after CRS-HIPEC for peritoneal metastasis in colorectal cancer (a phase 1 study). Front Med (Lausanne). 2023 Mar 1;10:1070362. doi: 10.3389/fmed.2023.1070362. eCollection 2023. PMID 36936230